CLINICAL TRIAL: NCT03628950
Title: The Analgesic Efficacy and Hemi-diaphragmatic Paralysis Assessment of Combined Infraclavicular-suprascapular Nerve Blocks Versus Standard Interscalene Brachial Plexus Block for Arthroscopic Rotator Cuff Repair
Brief Title: Interscalene Versus Combined Infraclavicular-suprascapular Nerve Blocks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Hany M Yassin, MD, Associate Professor of Anesthesiology, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: D165
Record Dates: First submitted 2018-07-21; First posted 2018-08-14 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain
Keywords: Interscalene block; Postoperative analgesia; Suprascapular nerve block; Infraclavicular nerve block; Arthroscopic rotator cuff repair; Hemi-diaphragmatic paralysis
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICSSB group (Active Comparator): infraclavicular suprascapular nerve block administered group
  Interventions: Procedure: ICSSB group
- ISB group (Active Comparator): interscalene nerve block administered group
  Interventions: Procedure: ISB group

INTERVENTIONS:
Procedure: ICSSB group — At supine position with abducted limb, the probe of ultrasound will be translocated in costoclavicular space; the subclavian artery will be identified. The three cords of the brachial plexus will be visualized lateral to the artery. By using an in-plane technique and a cephalad-to-caudate direction, the block needle will be advanced until its tip will be in the middle of three cords and 10 mL of 0.25 % bupivacaine Hydrochloride will be injected. Then at lateral decubitus position, by using in-plane technique the probe will be translocated in suprascapular fossa, lateral-to-medial direction, the block needle will be advanced until its tip in the floor of the suprascapular fossa ventral to the fascia of the supraspinatus muscle and 10 mL of 0.25 % bupivacaine Hydrochloride will be injected .
  Other Names: Infraclavicular suprascapular block group
  Arms: ICSSB group
Procedure: ISB group — The probe of ultrasound will be applied in lateral side of the neck at the level of the cricoid cartilage to obtain a view of the three hypoechoic structures which represent the roots of the brachial plexus. Using an in-plane technique and a lateral to-medial direction, the block needle will be advanced until its tip will be positioned under the prevertebral fascia between the two most superficial hypoechoic structures and 10 mL of 0.25 % bupivacaine Hydrochloride will be injected at level of C5-6 and another 10 ml of 0.25 % bupivacaine Hydrochloride will be injected at level of C7-8.
  Other Names: Interscalene group
  Arms: ISB group

SUMMARY:
The aim of this trial is to compare the analgesic efficiency and hemi-diaphragmatic paralysis of the standard ultrasound-guided interscalene (ISB) brachial plexus block with the combined use of costoclavicular approach of infraclavicular brachial plexus block and suprascapular nerve block (ICB-SSB) for patients undergoing arthroscopic rotator cuff repair.

Authors hypothesize that the combined use of ICB-SSB could lead to equivalent postoperative analgesic effect to the standard ISB with less hemi-diaphragmatic paralysis.

DETAILED DESCRIPTION:
The interscalene block main hindrance is the high risk of ipsilateral phrenic nerve block with sequential hemi-diaphragmatic paralysis.The combined use of conventional paracoracoid infraclavicular block (ICB) and suprascapular block (SSB) was not equivalent to the standard ISB regarding the analgesic efficacy , but has no hemi-diaphragmatic affection for patients undergone shoulder arthroscopic procedures.ICB can be achieved by another approach (costoclavicular) which blocks the brachial plexus at the mid infraclavicular fossa The patients scheduled for an elective arthroscopic rotator cuff repair will be randomly allocated by a computer-gener¬ated table into one of two study groups. The randomization sequence will be concealed in opaque sealed envelopes. The envelopes will be opened by the study investigators just after recruitments and admission to the operation room. Only assessors and data collectors will be blinded to the groups allocations.

Preoperative preparation:

Preoperative investigations will be done according to the local protocol designed to evaluate the patients. It includes complete blood count, blood sugar level, serum urea and creatinine, liver function tests, coagulation profile and electrocardiogram (ECG).

Intraoperative Management of Patients:

After arrival to the induction room, a 20G intravenous catheter will be placed in the upper limb opposite to the surgical site, and intravenous premedication (midazolam 2 mg and fentanyl 50 µg) will be administered to all patients. Supplemental oxygen (nasal cannulae at 2 Lmin-1), standard ASA monitoring (5-lead ECG, noninvasive blood pressure (NIBP), and pulse oximetry) will be applied throughout the procedure. All blocks will be performed under real-time ultrasound guidance (Philips clear vue350, Philips healthcare, Andover MA01810, USA).

The patients in both groups will initially receive superficial cervical plexus block. The block will be performed in supine position with the patients' head turned to the other side. Once the skin is appropriately cleaned and prepared with anti-septic, the high frequency linear array transducer (8-15 megahertz) will be placed over the lateral side of the neck at the midpoint of the posterior border of the sternocleidomastoid muscle(SCM). The transducer is positioned such that the tapering end (posterior border on the ultrasound image) of the SCM is in the center of the screen. The block needle (22-gauge, 50 mm, Stimuplex D®; B Braun, Germany) is then introduced from the posterior aspect through the skin and platysma and 10 ml of local anesthetic(LA) deposited just behind this landmark. Afterthat the patients will receive either ISB or ICB-SSB.

Following completion of the assessments of sensorimotor blocks at 30 min (see below), induction of general anesthesia will be achieved by intravenous propofol 1.5-2 mgkg-1, fentanyl 1 ugkg-1, and atracurium 0.5 mgkg-1. General anesthesia will be maintained by isoflurane 1.5 volume % in 2 lmin-1 oxygen-air mixture 50:50 and atracurium 0.1 mgkg-1 every 30 minutes. All subjects will be placed in the beach chair position slowly, and the surgical procedures will be completed by the same surgical team.

Intraoperatively, if the patient's heart rate or blood pressure exceeded 20% of the preoperative value, a 50-µg bolus dose of fentanyl will be administered. Deliberate hypotension technique will be used to keep systolic blood pressure at 90-100 mmHg range, mean blood pressure at 65-75 mmHg range, and heart rate at 60-70 bpm range by nitroglycerine intravenous infusion at a rate of 1-2 µgkg-1min-1. If excessive unwanted hypotension (systolic blood pressure less than 90 mmHg or mean blood pressure less than 65 mmHg) will be noted, 200 ml ringer acetate fluid bolus will be administered to regain the blood pressure to the desired range with reducing the infusion rate of nitroglycerine or stop it temporarily. Otherwise, 5 mg ephedrine increments will be used to secure save blood pressure readings range. Bradycardia (HR less than 50 bpm) will be corrected by atropine sulphate administration at a dose of 30 µg increments.

Assessment of Sensory and Motor Blockade:

* The extent of motor and sensory blockade will be evaluated by an anesthesiologist who will not be involved in the brachial plexus block 30 min after local anesthetics administration. Using an alcohol swab, the sensory blockade will be tested on the skin overlying the clavicle (supraclavicular nerves) and the lateral surface of the deltoid (axillary nerve). Each territory will be graded according to a three-point scale using a cold test: 0 = no block; 1 = analgesia (patient can feel touch, not cold); 2 = anesthesia (patient cannot feel touch).
* Motor function will be tested using shoulder abduction (axillary and suprascapular nerves) and external shoulder rotation (suprascapular nerve) according a three-point scale: 0 = no block; 1 = paresis; 2 = paralysis. blocks will be considered complete if, at 30 min, a global composite score six points (out of a maximum of eight points) will be achieved,5 incidence of complete block 30 minutes after injection will be recoded.

Assessment of hemi-diaphragmatic paralysis (HDP) using Ultrasound:

Ultrasound evaluation of the hemi-diaphragm will be assessed by a blinded trained radiologist. A low-frequency (2 to 5 MHz) curvilinear array transducer will be placed in the coronal plane at the midaxillary line to obtain an intercostal view. At the level of ribs eight to nine on the left and seven to eight on the right, the spleen or liver are centered with the rib shadows on either side. On deep inspiration, caudal descent of the liver or spleen precedes descent of the bright pleural line. The transducer will then be moved in both caudal and cephalad directions to visualize the end-inspiratory and end-expiratory levels of the pleural line, respectively, which will be then marked on the patient's skin. This process will be repeated before, after the chosen regional anesthetic technique and after recovery from general anesthesia in post-anesthetic care unit (PACU) with the patient in the same position. Minimal change signifies no block, but a reduction in this distance represents phrenic nerve block.

Postoperative Evaluation:

After completion of the surgical procedure, the patients extubated after fulfilment of the extubation criteria and then will be transferred to PACU for 2 h assessment. At PACU all patients will receive ketoprofen 100 mg and acetaminophen 1 gram by intravenous infusion over 30 min. Postoperative pain will be rated on a numerical scale ranging (NRS) from 0 (no pain) to 10 (worst imaginable pain) at 1-hr at PACU then at 4, 8, 12, and 24 hours postoperatively. The patients discharged to ward after fulfilment of discharge criteria and modified Aldrete score ≥9. ketoprofen 100 mg/12 h and acetaminophen 1 gram/8 h by intravenous infusion over 30 min will be continued for 48 h as parts of the postoperative pain control policy of the institution. Assessment of postoperative analgesia duration by recording the time of first request of analgesia. The duration of anesthesia time (defined as the time between the end of the local anesthetic injection for brachial plexus block and the postoperative administration of analgesic agents) will be recorded. Patients with NRS>5 will receive morphine sulphate IV at a bolus dose of 2-5 mg increments with maximum dose of 20 mg at 4 hours or 40 mg at 24 hours. Cumulative and interval amount of morphine consumption in 24 h will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* American Society association (ASA) physical status I to III patients who will be scheduled for an elective arthroscopic rotator cuff repair.

Exclusion Criteria

* Patient refusal
* preexisting (obstructive or restrictive) pulmonary disease or low baseline oxygen saturation
* contraindication to regional anesthesia (coagulopathy, allergy to local anesthetic, sever thrombocytopenia, pre-existing neuropathy in operative limb, infection at puncture site).
* sepsis
* hepatic or renal dysfunction.
* Advanced cardiovascular diseases
* chronic pain condition requiring the intake of opioids at home.
* prior surgery in the neck or infraclavicular/suprascapular fossa.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
The cumulative morphine consumption at first 24 hours postoperatively. | 24 hours after recovery from general anesthesia
  in milligram

SECONDARY OUTCOMES:
Assessment of hemidiaphragmatic paralysis | 5 minutes before intervention
  By using abdominal ultrasonography examination
Assessment of hemidiaphragmatic paralysis | 5 minutes after intervention
  By using abdominal ultrasonography examination
Assessment of hemidiaphragmatic paralysis by abdominal ultrasound examination | 10 minutes after recovery from general anesthesia
  By using abdominal ultrasonography examination
Assessment of postoperative pain | 1 hour after recovery from general anesthesia
  using numerical rate scale (NRS)(where 0=no headache and 10 = worst imaginable headache )
Assessment of postoperative pain | 4 hours after recovery from general anesthesia
  using numerical rate scale (NRS)(where 0=no headache and 10 = worst imaginable headache )
Assessment of postoperative pain | 8 hours after recovery from general anesthesia
  using numerical rate scale (NRS)(where 0=no headache and 10 = worst imaginable headache )
Assessment of postoperative pain | 12 hours after recovery from general anesthesia
  using numerical rate scale (NRS)(where 0=no headache and 10 = worst imaginable headache )
Assessment of postoperative pain | 24 hours after recovery from general anesthesia
  using numerical rate scale (NRS)(where 0=no headache and 10 = worst imaginable headache )
Assessment of postoperative pain | 48 hours after recovery from general anesthesia
  using numerical rate scale (NRS)(where 0=no headache and 10 = worst imaginable headache )
Interval morphine consumption dose | at 2 hours after recovery from general anesthesia
  in milligram
Interval morphine consumption dose | at 4 hours after recovery from general anesthesia
  in milligram
Interval morphine consumption dose | at 8 hours after recovery from general anesthesia
  in milligram
Interval morphine consumption dose | at 12 hours after recovery from general anesthesia
  in milligram
Interval morphine consumption dose | at 24 hours after recovery from general anesthesia
  in milligram
Interval morphine consumption dose | at 48 hours after recovery from general anesthesia
  in milligram
Incidence of complete sensory block | 30 minutes after end of local anesthetic injection
  using alcohol swab according to three point scale where 0= no block 1=analgesia (patient can feel touch not cold) 2=anesthesia (patient cannot feel touch)
Incidence of complete motor block | 30 minutes after end of local anesthetic injection
  using shoulder abduction and external rotation according to three point scale where 0= no block 1=paresis 2=paralysis
Intraoperative fentanyl dose consumption | At the end of surgical procedure
  In microgram
Incidence of nausea | 24 hours postoperative
  Opioid-related side effect
Incidence of vomiting | 24 hours postoperative
  Opioid-related side effect
Incidence of pruritus | 24 hours postoperative
  Opioid-related side effect
Incidence of excessive sedation | 24 hours postoperative
  Opioid-related side effect
Incidence of respiratory depression | 24 hours postoperative
  Opioid-related side effect
Incidence of urine retention | 24 hours postoperative
  Opioid-related side effect
time to first rescue analgesia | from recovery of general anesthesia up to 24 hours postoperativly
  in minutes
duration of the surgical procedure | At the end of surgical procedure
  in minutes
performance time of the intervention | 1 minute immediately after end of local anesthetic injection
  time from skin disinfection until the end of local anesthetic injection
Incidence of vascular puncture | within 3 seconds during performance of the blocks
  potential adverse events from intervention
Incidence of local anesthetic toxicity | 30 minutes after performance of the blocks.
  potential adverse events from intervention
Incidence of paresthesia | within 1 second during performance of the blocks
  potential adverse events from intervention
Incidence of Horner syndrome | 30 minutes after performance of the blocks.
  potential adverse events from intervention
Incidence of hoarseness of voice | 30 minutes after performance of the blocks.
  potential adverse events from intervention
Age | 6 hours before intervention
  in years
weight | 6 hours before intervention
  in kilogram(kg)
height | 6 hours before intervention
  in meters(m)
body mass index | 6 hours before intervention
  in kg/m square
Assessment of patients' satisfaction score for postoperative analgesia | after 72 hours postoperative
  poor=0; fair=1; good=2; excellent=3
Assessment of surgeon's' satisfaction score | At the end of surgical procedure
  poor=0; fair=1; good=2; excellent=3

CONTACTS AND LOCATIONS:
Overall Officials: Safaa G Ragab, MD, Study Director — Faculty of medicine, Fayoum university; Mohamed M Arafa, MD, Study Director — Faculty of medicine, Fayoum university
Locations (1):
- Fayoum University hospital, El Fayoum Qesm, Faiyum Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ullah H, Samad K, Khan FA. Continuous interscalene brachial plexus block versus parenteral analgesia for postoperative pain relief after major shoulder surgery. Cochrane Database Syst Rev. 2014 Feb 4;2014(2):CD007080. doi: 10.1002/14651858.CD007080.pub2. PMID 24492959
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Aliste J, Bravo D, Finlayson RJ, Tran DQ. A randomized comparison between interscalene and combined infraclavicular-suprascapular blocks for arthroscopic shoulder surgery. Can J Anaesth. 2018 Mar;65(3):280-287. doi: 10.1007/s12630-017-1048-0. Epub 2017 Dec 19. PMID 29270914
- [Background] Tran DQ, Elgueta MF, Aliste J, Finlayson RJ. Diaphragm-Sparing Nerve Blocks for Shoulder Surgery. Reg Anesth Pain Med. 2017 Jan/Feb;42(1):32-38. doi: 10.1097/AAP.0000000000000529. PMID 27941477
- [Background] Karmakar MK, Sala-Blanch X, Songthamwat B, Tsui BC. Benefits of the costoclavicular space for ultrasound-guided infraclavicular brachial plexus block: description of a costoclavicular approach. Reg Anesth Pain Med. 2015 May-Jun;40(3):287-8. doi: 10.1097/AAP.0000000000000232. No abstract available. PMID 25899958